CLINICAL TRIAL: NCT06997796
Title: Sprayed-In Medicated Powder for Less-Invasive Epistaxis Treatment Using Tranexamic Acid: The Bloody SIMPLE Treatment Pilot Study
Brief Title: Treatment of Nosebleeds in the Emergency Department With Powder Tranexamic Acid
Acronym: Bloody SIMPLE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dr. Anne Conlin (Other)
Collaborators: University of Ottawa (Other)
Responsible Party: Sponsor-Investigator, Dr. Anne Conlin, Peterborough Regional Health Center Staff Otolaryngologist-Head & Neck Surgeon; Assistant Professor University of Ottawa, Peterborough Regional Health Centre
Organization: Peterborough Regional Health Centre (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2025-05-13; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Epistaxis Nosebleed
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tranexamic acid powder applied intranasally (Experimental)
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — Tranexamic acid powder intranasally

SUMMARY:
Nosebleeds are very common, occurring in 60% of the population; in some patients, nosebleeds are a life-threatening emergency. To stop a nosebleed in the emergency department, doctors usually have to burn the nose (called cauterization) or insert pledgets (called nasal packing) into the nose to apply direct pressure to the bleeding site. Nasal packing can cause pain and discomfort at the time it is inserted in the nose and again when it is removed. In rare cases it can cause a range of complications: minor complications include scar bands in the nose, but serious complications of nasal packing have also occurred, including death. Nasal packing can also present risks to doctors, such as the risk of contracting airborne and bloodborne infections, like COVID-19 and HIV.

Tranexamic acid in pill form or given directly into a vein is a medication that is currently used for nosebleeds. This study looks to evaluate if tranexamic acid in powder form sprayed directly in the nose can be used as an alternative to cauterization or nasal packing for the treatment of nosebleeds.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Adults 18 years or older
* Male or female
* Presenting to the ED with active, spontaneous epistaxis. Anterior versus posterior epistaxis will be identified a priori. Anterior epistaxis is operationally defined as active nasal bleeding that occurs anterior to the anterior limit of the middle turbinate, visible by anterior rhinoscopy.

Exclusion Criteria:

* Prior sinonasal surgery within the preceding 1 month.
* Patients who required medical treatment for epistaxis in the preceding 30 days.
* Septum perforation.
* Known history of bleeding disorders, including thrombocytopenia, hemophilia, hereditary hemorrhagic telangiectasia, or von Willebrand disease.
* History of known thromboembolic disease, including subarachnoid hemorrhage, stroke, or TIA.
* Known history of disease of the central nervous system, including seizures, convulsions, or intra-cerebral disease processes/lesions.
* Known or suspected history of significant skull base trauma, including skull base fracture or cerebrospinal fluid leak.
* Known history of acquired disturbances of colour vision.
* Known hematuria or any bleeding related to the kidney.
* Pregnant and/or lactating women.
* History of known allergy or sensitivity to the study medication.
* Presence of signs or symptoms of concomitant emergent conditions, including myocardial infarction, stroke, major trauma, shock, or hemodynamic instability.
* Patients with other medical conditions including cognitive limitations or impairment due to substance abuse.
* Patients with any other condition that, in the opinion of the investigator, may present an unreasonable risk to the patient, may make the patient unreliable, or may interfere with the study assessments.
* Current participation in another interventional clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Cessation of epistaxis | Day 1
  Number of participants for whom epistaxis ceased after treatment

SECONDARY OUTCOMES:
Time to cessation of epistaxis | Day 1
  Measured in minutes
Pain of the treatment | Day 1
  Participants' perception of pain will be measured using the Visual Analog Scale (VAS), ranging from 0 (no pain) to 10 (worst pain possible).
Total time in the Emergency Department | Day 1
  Measured in minutes
Number of participants who returned to the Emergency Department for treatment of epistaxis | within the first 24 hours and the first 5 days after treatment

OTHER OUTCOMES:
Age | Day 1
Anticoagulant and/or antiplatelet medication use | Day 1
Type of epistaxis | Day 1
  Anterior versus posterior epistaxis
Adverse events and/or patient-reported side effects | up to 3 weeks
Treatment site complications | up to 3 weeks
  Participants will be examined for complications, including synechiae or nasal infections

CONTACTS AND LOCATIONS:
Overall Officials: Anne Conlin, Assistant Professor, University of Ottawa, HBA&Sc, MD, FRCSC, Principal Investigator — Peterborough Regional Health Center; University of Ottawa
Locations (1):
- Peterborough Regional Health Centre, Peterborough, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes